CLINICAL TRIAL: NCT02587988
Title: A Randomized, Double-blind, Multicenter, Phase Ⅲ Study to Evaluate the Efficacy and Safety of HCP1302 in Both Erectile Dysfunction and Hypertension Patients Being Treated With HGP0904
Brief Title: Trial to Evaluate the Efficacy and Safety of HCP1302
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-TARO-301
Record Dates: First submitted 2015-10-25; First posted 2015-10-27 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Erectile Dysfunction; Hypertension
Keywords: Erectile dysfunction & Hypertension
MeSH Terms: conditions — Erectile Dysfunction; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCP1302+HGP0904Placebo (Experimental): HCP1302+HGP0904Placebo for 12weeks
  Interventions: Drug: HCP1302; Drug: Placebo (for HGP0904)
- HCP1302Placebo+HGP0904 (Active Comparator): HCP1302Placebo+HGP0904 for 12weeks
  Interventions: Drug: HGP0904; Drug: Placebo (for HCP1302)

INTERVENTIONS:
Drug: HCP1302
  Arms: HCP1302+HGP0904Placebo
Drug: HGP0904
  Arms: HCP1302Placebo+HGP0904
Drug: Placebo (for HCP1302)
  Arms: HCP1302Placebo+HGP0904
Drug: Placebo (for HGP0904)
  Arms: HCP1302+HGP0904Placebo

SUMMARY:
Trial to Evaluate the Efficacy and Safety of HCP1302

DETAILED DESCRIPTION:
A Randomized, Double-blind, Multicenter, Phase Ⅲ study to Evaluate the Efficacy and Safety of HCP1302 in Both Erectile Dysfunction and Hypertension Patients being Treated with HGP0904

ELIGIBILITY:
At Visit1

1. ≥19 age
2. Hypertension Patients who need amlodipine 5mg
3. Abnormal Erectile function ≥ at least 3months based on screening date
4. Patients who are expected to frequent use of Tadalafil (at least two times for weeks)
5. Patients understood the consents and purpose of this trial and signed informed consent form

At Visit2

1. 90≤ sitSBP < 140 mmHg and 50 ≤ sitDBP < 90 mmHg
2. Sexual dysfunction rate ≥ 50% for 4 weeks run-in period
3. International Index of Erectile Function(IIEF)- Erectile Function(EF) domain score ≤ 25

Exclusion Criteria:

1. History of hypersensitivity to Amlodipine or Tadalafil
2. Has a severe liver disorder(Child-Pugh Class C) or liver enzyme (AST, ALT) level exceeds 3 times more than normal upper range
3. Has a clinically significant renal failure (Scr > 2mg/dl)
4. Uncontrolled diabetes mellitus (HbA1C >12%)
5. At screening date, blood pressure gap of selected arms is sitSBP ≥20mmHg or sitDBP ≥10mmHg
6. Taking PDE-5 inhibitors or other therapeutic agents for Erectile Dysfunction within 7 days based on screening date
7. No reaction to PDE-5 inhibitors

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2014-09; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change of IIEF-EF domain score | baseline and 12 weeks
Change of sitting diastolic blood pressure | baseline and 12 weeks

SECONDARY OUTCOMES:
Change of sitting diastolic blood pressure | baseline, 4weeks and 8weeks
Change of sitting systolic blood pressure | baseline,4weeks, 8weeks and 12 weeks
Change of IIEF-EF domain score | baseline, 4weeks and 8weeks

IPD SHARING:
Plan to Share IPD: No